CLINICAL TRIAL: NCT00521170
Title: Randomized, Monocenter, Double Blind, Placebo-controlled, Single Oral Dose, Three-way Cross Over Study, to Compare Levocetirizine and Desloratadine on Allergen-induced Wheal and Flare Reaction During 24 Hours in 18 Adult Allergic Volunteers.
Brief Title: Wheal and Flare Reaction During 24 Hours in Allergic Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A00373; Eudract Number: 2004-001089-41
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2009-09

CONDITIONS: Allergy
Keywords: Levocetirizine; Wheal and flare; Allergic
MeSH Terms: conditions — Hypersensitivity; Urticaria | interventions — levocetirizine

INTERVENTIONS:
Drug: Levocetirizine

SUMMARY:
Compare the activity of 5 mg levocetirizine and 5 mg desloratadine on allergen-induced wheal and flare reaction.

ELIGIBILITY:
Inclusion Criteria:

* Male and female allergic volunteers: Diagnosed allergy based on medical history and on positivity to skin tests to at least one of the standardized allergen including grass pollens, tree pollens, house dust mites, cat and dog dander and with a positive RAST for the specific selected allergen ≥ class 2

Exclusion Criteria:

* Pregnancy or lactating females, or females with childbearing potential without reliable contraception
* History or presence of any chronic or acute illness or disorder capable of altering the absorption, metabolism or elimination of drugs, or constituting a risk factor when taking the trial medication
* Heavy caffeine drinker (> 5 cups of coffee, tea, cola, etc … per day)
* Any drug treatment, including prescribed or non-prescription medicines (except hormonal contraceptives or post-menopausal hormonal replacement therapy for females and occasional use of paracetamol not exceeding 2 g/day with a maximum dose of 10 g per 14 days), taken from 14 days before study drug administration; the wash-out period after intake of systemic corticosteroids is at least 4 weeks
* Known allergy/intolerance to the study drug or any medicine chemically related to study drug or its excipients (lactose, cellulose...)
* Participation in another clinical trial, blood donation or significant blood loss (> 450 mL) less than 12 weeks before the study drug administration
* Skin irritant or 48 hours UV exposure before each visit
* Immunotherapy received during the current year
* Any clinical conditions that, in the opinion of the Investigator, would make the subject unsuitable for the trial

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Dates: Start 2004-11; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Compare the activity of levocetirizine and desloratadine on allergen-induced wheal and flare reaction. Response to allergen administered by skin prick test (SPT) measured by the wheal and flare surface areas | 15 minutes

SECONDARY OUTCOMES:
Compare the AUC from pre-dose to 24 hours post-dose between levocetirizine and placebo and between desloratadine and placebo obtained for wheal and for flare areas. Compare the AUC from pre-dose to 12 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (2):
- France (2):
  - Illkirch-Graffenstaden
  - Strasbourg